CLINICAL TRIAL: NCT04151147
Title: Effect of Concentrated Growth Factors on Frequency of Alveolar Osteitis Following Partially Erupted Mandibular Third Molar Surgery: A Randomized Controlled Clinical Study
Brief Title: Effect of CGF on Frequency of Alveolar Osteitis Following Partially Erupted Mandibular Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gözde Işık, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Oral Surgery
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Alveolar Osteitis; Impacted Tooth
Keywords: Third molar surgery; Alveolar osteitis; Platelet concentrates
MeSH Terms: conditions — Dry Socket; Tooth, Impacted | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGF application in the extraction socket (Experimental): Partially impacted third molar was extracted with the help of straight elevator and third molar forceps. After extraction, any remains of the dental follicle were removed and the extraction sockets were irrigated with 60 mL of sterile saline. CGF fibrin gel was then randomly placed into one socket and wound closure was completed with silk suture.
  Interventions: Procedure: Concentrated Growth Factor (Test group)
- non-CGF application in the extraction socket (Experimental): Opposite side of the patient was considered as the control. After extraction of the third molar, dental follicle were removed and to prevent the flap laceration, bone contouring was also performed under sterile saline irrigation. Finally, wound closure was completed with silk suture.
  Interventions: Procedure: Non-Concentrated Growth Factor (Control group)

INTERVENTIONS:
Procedure: Concentrated Growth Factor (Test group) — The patients' blood was collected in 9 ml glass tubes and immediately centrifuged to prevent coagulation in special centrifuge device. The CGF program was set up as follows: accelerated for 30 seconds so as to reach 2700 rpm, rotated for 2 minutes, then reduced to 2400 rpm, then rotated again for 4 minutes and accelerated to 2700 rpm, rotated for 4 minutes, then accelerated to 3000 rpm for 3 minutes, and decelerated for 36 seconds to stop. The middle layer in the tube was separated by the ''Buffy coat'' containing the CGFs fibrin gel using forceps and scissor. Then, this fibrin gel was inserted in the extraction cavity.
  Arms: CGF application in the extraction socket
Procedure: Non-Concentrated Growth Factor (Control group) — Third molar extraction was performed under local anesthesia. Following the extraction, the socket was sutured and natural healing process was observed. This side was considered as a control group.
  Arms: non-CGF application in the extraction socket

SUMMARY:
The aim of this prospective study was to assess the effectiveness of concentrated growth factors (CGFs) in preventing the development of alveolar osteitis (AO) after the extraction of partially-erupted mandibular third molars.

This study was designed as a randomized controlled clinical trial. In each case, one socket received CGFs and the other served as a control. The predictor variable was the CGFs application and the sides were categorized as 'CGFs' and 'non-CGFs'. The outcome variable was the development of AO during the first postoperative week. Also, demographic variable included age and gender was noted.

DETAILED DESCRIPTION:
The investigators designed and implemented a randomized single-blind clinical trial.Randomization was performed by simple coin toss to select the side of CGFs fibrin gel placement before the commencement of third molar surgery. In this way, the sides in each patient were randomly divided into 2 study groups:

Group I (test) - with CGFs placed in the extraction socket Group II (control) - without CGFs placement All operations were performed under local anesthesia by the same surgeon. An envelope flap was raised to provide access. Bone removal was done with the help of stainless steel burs. Constant irrigation with saline was used while removing bone to prevent thermal necrosis. Third molar was luxated with the help of straight elevator and then extracted with the help of third molar forceps. After extraction, any remains of the dental follicle were removed and the extraction sockets were irrigated with 60 mL of sterile saline. To prevent the flap laceration, bone contouring was also performed under sterile saline irrigation. CGFs fibrin gel was then randomly placed into one socket and the opposite side was considered as the control. Finally, wound closure was completed with silk suture.

The primary outcome variable was AO, classified as present or absent.It is characterized by postoperative pain in and around the extraction side, which increases in severity within first week after the extraction, accompanied by a partially or totally disintegrated blood clot within the alveolar socket, with or without halitosis. Other defining symptoms that have been reported in the literature are radiating pain towards the temporal region and ear, inflamed gingival margin, ipsilateral regional lymphadenopathy and, less commonly, low-grade fever.

ELIGIBILITY:
Inclusion Criteria:

* Patients Age ≥ 18 years of age
* Willing and able to provide informed consent
* Ability to cooperate with the requirements of the study protocol
* Healthy patients without medical diseases or a history of bleeding problems
* Patients with the need of extraction of third molars
* The third molars had to be symmetrical, partially-erupted and in the Class I, Level B according to Pell & Gregory classification and in the vertical angulations according to Winter's classification.

Exclusion Criteria:

* Patients who have pre-existing abscess or cellulitis, acute pericoronitis, or pre-existing conditions such as an odontogenic cyst or tumour associated with their third molars
* Patients who were pregnant and breastfeeding
* Patients with drug usage such as bisphosphonate, steroids and antidepressants
* Patients who had a smoking habit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Presence of alveolar osteitis formation | Change of alveolar osteitis formation at 7 days.
  Clinical data was collected with regard to alveolar osteitis formation on the 3rd and 7th days after surgery with the following characteristics: 1) progressive and severe pain in and around the extraction side within first week; 2) partially or totally loss of blood clot and exposure of the alveolar bone with or without halitosis. Patients who met one of the criterias, were taken to be alveolar osteitis.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Özveri Koyuncu, Study Director — Ege University
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozveri Koyuncu B, Isik G, Ozden Yuce M, Gunbay S, Gunbay T. Effect of concentrated growth factors on frequency of alveolar Osteitis following partially-erupted mandibular third molar surgery: a randomized controlled clinical study. BMC Oral Health. 2020 Aug 17;20(1):222. doi: 10.1186/s12903-020-01210-7. PMID 32807173